CLINICAL TRIAL: NCT06575569
Title: Effect of High-intensity Intermittent Rehabilitation Training on Cardiopulmonary Function After PCI in Patients With Coronary Heart Disease
Brief Title: Effect of HIIT on Cardiopulmonary Function After PCI in Patients With Coronary Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Chen Leilei, Director, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIIT-PCI
Record Dates: First submitted 2024-08-20; First posted 2024-08-28 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high-intensity interval training (HIIT) group (Experimental): intensive interval training under the care of specialists for 12 weeks, 30-40 minutes per week, including starting 5-minute warm-up and last 5-minute cooling-off period, during exercise including 4 intervals, 85-95% of maximum heart rate (HR) reserve for 4 minutes, followed by 50-70% of maximum HR reserve for 3 minutes, so cycling 4 times.
  Interventions: Behavioral: high-intensity interval training
- Moderate-intensity continuous training (MCT) group (Active Comparator): patients exercise prescription for 12 weeks, 30-40 minutes, including 5 minutes of warm-up and cooling-off period of the last 5 minutes, during exercise intensity is 70-75% maximum heart rate reserve. The warm-up and cooling-off periods can be performed by stretching, flexibility exercises (i. e., neck, shoulders, upper back, hips, and ankles), and medium to low intensity (50-70% heart rate reserve).
  Interventions: Behavioral: Moderate-intensity continuous training

INTERVENTIONS:
Behavioral: high-intensity interval training — Patients had no adverse events after 2 weeks of adaptive exercise training and voluntarily continued participants, intensive interval training under the care of specialists for 12 weeks, 30-40 minutes per week, including starting 5-minute warm-up and last 5-minute cooling-off period, during exercise including 4 intervals, 85-95% of maximum heart rate (HR) reserve for 4 minutes, followed by 50-70% of maximum HR reserve for 3 minutes, so cycling 4 times. Specific exercise logs will be issued for patients to record exercise conditions and related exercise data, encouraged to exercise regularly and health education materials pushed by cardiovascular nurses.
  Other Names: HIIT
  Arms: high-intensity interval training (HIIT) group
Behavioral: Moderate-intensity continuous training — Using routine postoperative care and follow-up, establish WeChat group as contact for postoperative follow-up, no adverse events after 2 weeks of adaptive exercise training and voluntary participants, patients exercise prescription for 12 weeks, 30-40 minutes, including 5 minutes of warm-up and cooling-off period of the last 5 minutes, during exercise intensity is 70-75% maximum heart rate reserve. The warm-up and cooling-off periods can be performed by stretching, flexibility exercises (i. e., neck, shoulders, upper back, hips, and ankles), and medium to low intensity (50-70% heart rate reserve). Specific exercise logs will be issued for patients to record exercise conditions and related exercise data, encouraged to exercise regularly and pushed health education materials by cardiovascular nurses.
  Other Names: MCT
  Arms: Moderate-intensity continuous training (MCT) group

SUMMARY:
Both the gut microbiome and exercise are closely related to human health, but the understanding of the effect of high-intensity interval training (HIIT) on cardiopulmonary function and human intestinal flora is still further study.

DETAILED DESCRIPTION:
As one of the most causes mortality all over the world, coronary heart disease (CHD) contributes to about 1.78 billion in Europe, 0.36 all deaths in the United States and over 110 million individuals worldwide each year, which has been a heavy burden on health expenditure. The treatment ways of CHD mainly include life way, drugs, and percutaneous coronary intervention (PCI). Even though, in past decades PCI technique has developed rapidly and today is a main treatment for patients with CHD. It was reported than healthcare costs will reach $177 billion by 2024 in the United States. In Europe, productivity losses were £13,953 per person per year because of CHD. Despite the traditional treatment, costs and mortality owing to CHD are still high, which highlights the need for research of the relationships between CHD and systems other than the cardiovascular system and comorbidities. The investigators need to search for new measures to improve traditional treatment ways of CHD. With the development of high-throughput sequencing technology, numbers of studies have showed that closely relationship between gut microbiota and cardiopulmonary function, blood glucose, lipid and cholesterol profiles and some inflammatory markers in patients with chronic disease. Regulation of intestinal flora may have preventive effect on disease. However, the study for relationship of CHD and gut microbiota is few reports. Health is a topic of common concern around the world. Increasing attention to the status of CHD and finding exercise prescriptions that effectively regulate the intestinal flora may lay the foundation for the prevention and treatment of chronic diseases such as CHD.

Some experiments have demonstrated that High-intensity interval training (HIIT) can change the diversity and metabolic capacity of gut microbiota. Therefore, it is necessary to conduct more studies to figure out whether exercise training could improve gut microbiota and bring benefit to human.

This study will explore whether 12 weeks of HIIT can effectively change the structure of human with CHD intestinal flora, so as to provide a theoretical basis for the human with CHD and exercise intervention in the treatment of intestinal flora related diseases.

ELIGIBILITY:
Inclusion Criteria:

* coronary angiography confirmed patients with coronary heart disease, which was at least one coronary vessel with a stenosis greater than 70%.
* Age is 18-70 years old, and the clinical sinus rhythm is stable.
* Left ventricular ejection fraction was> 40%.
* Informed consent and voluntary participation.

Exclusion Criteria:

* Patients with severe organic cardiac and lung diseases.
* Patients with hemiplegia and other physical action disorders.
* A history of mental illness.(4) Uncontrolled hypertension, and hemodynamic instability.
* Severe nephropathy and severe peripheral artery disease.
* Patients with bone and joint diseases who are not suitable for exercise.
* Uncontrolled endocrine system and other diseases.
* Antibiotics and anti-diarrheal medications have not been used for at least 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2023-06-17 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Gut microbiome | 12 weeks
  Fecal DNA isolation was performed using the QIA amp Fast DNA Stool Mini Kit. After DNA extraction, fecal DNA was used for library preparation, and whole-genome shotgun sequencing was performed on the Illumina NovaSeq-6000 plat- form. From the raw metagenomic sequencing data, low-quality reads were discarded by the sequencing facility, and reads belonging to human contaminations were removed by mapping the data to the reference genomes using Bowtie2 (RRID:SCR _ 016368 ; v2.4.5). After filtering, on average, 54.8 million (SD = 14.7 million) paired reads per sample were obtained for subsequent analysis.
Plasma metabolite Traumatic acid | 12 weeks
  Plasma
6MWT | 12 weeks
  6-minute walk test
VO2peak | 12 weeks
  CPET

CONTACTS AND LOCATIONS:
Overall Officials: Leilei Chen, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Department of Cardiology ,the First Affiliated Hospital of Nanjing Medical University, Nanjing, China

IPD SHARING:
Plan to Share IPD: No